CLINICAL TRIAL: NCT03327493
Title: Impact of Adrenoreceptor Expressions on Inflammatory Pattern in Refractory Cardiogenic Shock Patients Treated by Veno-arterial Extra-Corporeal Membrane Oxygenation
Brief Title: Impact of Adrenoreceptor Expressions on Inflammatory Pattern in Refractory Cardiogenic Shock Under VA ECMO
Acronym: ADRECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Dr Antoine KIMMOUN, PU-PH, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00707-44
Record Dates: First submitted 2017-09-21; First posted 2017-10-31 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Shock, Cardiogenic; Extra-Corporeal-Life-Support ( ECLS); Autonomic Nervous System Diseases; Inflammation
Keywords: Cardiogenic shock; Extra-Corporeal-Life-Support (ECLS); inflammation; adrenergic system
MeSH Terms: conditions — Shock, Cardiogenic; Autonomic Nervous System Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Refractory cardiogenic shock patients under ECLS. Assessment at ECLS start, day 3 and Day "ECLS weaning" for various biological variables
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory cardiogenic shock under ECLS (Other)
  Interventions: Diagnostic Test: Biological

INTERVENTIONS:
Diagnostic Test: Biological — We will assess in all patients under ECLS for the treatment of a cardiogenic shock at day 0 (ECLS initiation) day 3 and day "ECLS weaning" :
  Biological assessment:
  1. Adrenoreceptors α1, α2, β1, β2, β3 on monocytes and lymphocytes T helper by flow cytometry
  2. Lymphocytes Th1/Th2 pattern by flow cytometry
  3. Cytokines on plasma : Interleukin (IL) 4, IL 12, TNF α, INF γ , IL1, IL6, IL10
  Clinical assessment:
  1. Hemodynamic parameters
  2. Cumulated doses of catecholamines
  3. Cardiac output variation measured by echocardiography during a standardized weaning procedure of ECLS at a constant mean arterial pressure (only on day 3 and Day "ECLS weaning")

SUMMARY:
Refractory cardiogenic shock is characterized by a decreased in cardiac output with hypo-responsiveness to increasing doses of catecholamines resulting in a profound tissular ischemia. VAECMO, by restoring a circulatory flow, could be associated to a major reperfusion syndrome which may lead some patients to multiple organ failures and death. Pathophysiology of this syndrome includes 1/an hyper-adrenergic state secondary to the over activation of the sympathetic system and 2/ a major release of pro-inflammatory cytokines. As adrenoreceptors are also exhibited on immunes cells, the pro-inflammatory state might be enhanced by the over-activation of the sympathetic system.

DETAILED DESCRIPTION:
NB : A repartition according to other ongoing study (HYPOECMO NCTNCT02754193) is planned

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU
* Refractory cardiogenic shock

  * Cardiogenic shock: Systolic Arterial Pressure <90mmHg, or Mean Arterial Pressure <65mmHg, adequate volemia, peripheral hypoperfusion symptoms, cardiac index < 2.2 l/min/m2)
  * Refractory state: hypo responsiveness to norepinephrine AND/OR persisting profound hypo perfusion clinical symptoms despite optimal resuscitation
* needing an Extra-Corporeal-Life-Support
* informed consent from relatives or patient
* Affiliation to a social security regimen
* Preliminary medical examination

Exclusion Criteria:

* Patients under ECLS for a/an :

  * Cardiotoxic poisoning
* Human immunodeficient Virus or Viral hepatitis C
* Patient < 18 yo
* Pregnancy
* Patient under protective supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Cytokines (plasma TNF α, INF γ, IL4, IL 12, IL1 IL 6 IL 10) | day 0 (ECLS initiation), day 3, day "ECLS weaning"
  Exposition variable will be the density of α1, α2, β1, β2, β3-adrenoreceptors on immune cells (monocytes and lymphocytes T helper)

SECONDARY OUTCOMES:
Change in hemodynamic parameters | day 0 (ECLS initiation), day 3, day "ECLS weaning"
  Arterial pressures
Change in hemodynamic parameters | day 0 (ECLS initiation), day 3, day "ECLS weaning"
  heart rate
Change in hemodynamic parameters | day 0 (ECLS initiation), day 3, day "ECLS weaning"
  cumulated doses of catecholamines
Cardiac output variation during a weaning ECLS procedure | day 3, day "ECLS weaning"
  At a constant mean arterial pressure (65-75 mmHg), measurement by echocardiography of cardiac output at 2 times:
  * baseline (3L/min of ECLS flow)
  * after 45 min at weaning output (1.5 L/min of ECLS flow) Variation of norepinephrine doses will be also recorded
Mortality | 28 days and 90 days
Change in TH1 and TH2 pattern | day 0 (ECLS initation), day 3, day "ECLS weaning"
  Assessment in CD3/CD4 + cells of INF γ; IL12 (TH1) and IL4 (TH2)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Kimmoun, MD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No